CLINICAL TRIAL: NCT02847481
Title: A Pilot Study to Evaluate Fecal Microbiota Transplantation Engraftment in Irritable Bowel Syndrome
Brief Title: A Study to Evaluate Fecal Microbiota Transplantation Engraftment in IBS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: OpenBiome (Industry)
Responsible Party: Principal Investigator, Anthony Lembo, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P000211
Record Dates: First submitted 2016-07-12; First posted 2016-07-28 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation; myotrophin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- fecal microbiota transplantation (Experimental): fecal microbiota transplantation
  Interventions: Procedure: fecal microbiota transplantation
- placebo fecal microbiota transplantation (Placebo Comparator): placebo fecal microbiota transplantation
  Interventions: Drug: placebo fecal microbiota transplantation
- FMT after antibiotic pretreatment v1 (Experimental): fecal microbiota transplantation after antibiotic pretreatment
  Interventions: Procedure: fecal microbiota transplantation; Procedure: FMT with antibiotic pre-treatment (v1)
- FMT after antibiotic pretreatment v2 (Experimental): fecal microbiota transplantation after antibiotic pretreatment
  Interventions: Procedure: fecal microbiota transplantation; Procedure: FMT with antibiotic pre-treatment (v2)

INTERVENTIONS:
Procedure: fecal microbiota transplantation — fecal microbiota transplantation
  Arms: FMT after antibiotic pretreatment v1; FMT after antibiotic pretreatment v2; fecal microbiota transplantation
Drug: placebo fecal microbiota transplantation — placebo fecal microbiota transplantation
  Arms: placebo fecal microbiota transplantation
Procedure: FMT with antibiotic pre-treatment (v1) — FMT with antibiotic pre-treatment (v1)
  Arms: FMT after antibiotic pretreatment v1
Procedure: FMT with antibiotic pre-treatment (v2) — FMT with antibiotic pre-treatment (v2)
  Arms: FMT after antibiotic pretreatment v2

SUMMARY:
This is a randomized pilot study to characterize engraftment of a donor's microflora onto patients with Irritable Bowel Syndrome with diarrhea following fecal microbiota transplantation.

ELIGIBILITY:
Inclusion Criteria:

* IBS with diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
stable engraftment of donor microbiota | 10 weeks
  Stable engraftment will be defined with the Jensen-Shannon Divergence (JSD) between the bacteria community measured in the donor and recipient. Engraftment scores will be defined by the ratio between the JSD in comparison between the recipient and donor and the recipient and other healthy donors not providing material for their FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Singh P, Alm EJ, Kelley JM, Cheng V, Smith M, Kassam Z, Nee J, Iturrino J, Lembo A. Effect of antibiotic pretreatment on bacterial engraftment after Fecal Microbiota Transplant (FMT) in IBS-D. Gut Microbes. 2022 Jan-Dec;14(1):2020067. doi: 10.1080/19490976.2021.2020067. PMID 35014601